CLINICAL TRIAL: NCT05168345
Title: A Prospective Patient Education Program for IBD Patients - Impact on Patient Disease Understanding, Patient Reported Outcomes and Clinical Characteristics
Brief Title: A Prospective Patient Education Program for IBD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Eli Sprecher, MD, Director of clinical trails, Tel-Aviv Sourasky Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0285-18
Record Dates: First submitted 2020-06-11; First posted 2021-12-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Educational Course

STUDY DESIGN:
Intervention Model Description: Arm 1: IBD patients, patients of other chronic GI diseases' and healthy volunteers
  Both groups will be asked to fill in the "knowledge questionnaire" and the "self-assessment of knowledge questionnaire" once, during their routine visit to the GI department. Results of the questionnaire will be compared between the groups.
  IBD Patient's knowledge will also be subjectively assessed by their treating physician during their routine clinical visit, and knowledge scores will be compared (physician and questionnaire). Patients who will agree, will be asked to fill in the knowledge questionnaire a second time after two weeks for reliability testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IBD patients (Experimental): Arm 1: IBD patients, patients of other chronic GI disease' and healthy volunteers
  Both groups will be asked to fill in the "knowledge questionnaire" and the "self-assessment of knowledge questionnaire" once, during their routine visit to the GI department. Results of the questionnaire will be compared between the groups.
  IBD Patient's knowledge will also be subjectively assessed by their treating physician during their routine clinical visit, and knowledge scores will be compared (physician and questionnaire). Patients who will agree, will be asked to fill in the knowledge questionnaire a second time after two weeks for reliability testing. Patients will be recruited to represent all stages of diagnosis and all patient age groups. This will be done by recruitment of six main participant groups stratified by age (18-23 years, 24-36 years, 42-52 years, 53-70 years) and disease duration (<1 year since diagnosis, ≥1 year since diagnosis)
  Interventions: Other: Course and web information

INTERVENTIONS:
Other: Course and web information — The interventional phase of the study will be conducted on IBD patients only. Patients will undergo two interventional periods which will include:
  1. Self-selected information from the internet - patients will be asked to independently search the web for information regarding the categories of information which are discussed in the online course.
  2. An online, interactive IBD course. Lectures will be passed by the multidisciplinary team of the IBD Center which includes IBD gastroenterologists, an IBD nurse, an IBD dietitian, and a social worker.

SUMMARY:
During the past few decades, key medical organizations have highlighted the importance of patient education and support. Evidence suggests that improving inflammatory bowel disease (IBD) patients' knowledge of their disease may empower patients to use more adaptive coping strategies and compliance with therapy and medical follow-up. Medical knowledge of disease pathophysiology and treatment are important determinants of early stage self-management in newly diagnosed IBD patients, and of adherence to therapy. Level of patient knowledge has been associated with significantly lower health care costs, possibly through improving patients behavioral choices leading to improved long-term clinical outcomes (such as disease activity, hospitalization and surgeries) and through preventive medicine, such as vaccinations, and screening for cancer prevention.

Despite availability of multiple alternatives for raising disease education levels, many adolescent and adult patients consistently show low levels of comprehension of their disease state and treatment regimen. The primary aim of this study is to evaluate the effect of a video based educational program for IBD patients on patient knowledge and understanding of their disease, patient reported outcomes and quality of life.

DETAILED DESCRIPTION:
To evaluate the effect of a video based educational program for IBD patients on patient knowledge and understanding of their disease, patient reported outcomes and quality of life

Methods Study design: An open label, non-randomized clinical trial. Study population: IBD patients (n=140) will be recruited from the clinical setting of the IBD clinic within the Tel Aviv Medical Center (TLVMC) Gastrointestinal (GI) department. Patients will be recruited to represent all stages of diagnosis and all patient age groups. This will be done by recruitment of six main participant groups stratified by age (18-23 years, 24-36 years, 42-52 years, 53-70 years) and disease duration (<1 year since diagnosis, ≥1 year since diagnosis)

Inclusion criteria

1. Diagnosis of IBD and , other GI chronic diseases or healthy volunteers
2. Age 18-70 years
3. Minimal skills of computer and internet use

Exclusion criteria

1. Severe disease - malignant disease, hepatic failure, renal failure, cardiovascular, metabolic, neurological disease
2. Inability to sign an informed consent
3. Inability to complete the study protocol
4. For the intervention phase of the study, IBD patients will be excluded if they score high on the IBD knowledge questionnaire (>80%)

Withdrawal from the study

1. Inability to complete the study protocol

Methods Eligible patients will sign an informed consent form after being informed of the study protocol.

IBD knowledge questionnaire validation The validation process of the study questionnaire will be conducted on the entire study population.

Statistical analysis:

All statistical analyses will be performed using statistical software platform (SPSS) version 23.0 for Windows.

All patients that will be fully adhering to the study's protocol (considered as preforming ≥ 80% of exercises) will be included in data analysis. In addition, there will be intention-to-treat analysis that will include patients who will be excluded because of non-adherence to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IBD, GI chronic diseases or healthy volunteers
* Age 18-70 years
* Minimal skills of computer and internet use

Exclusion Criteria:

* Severe disease
* Inability to sign an informed consent
* Inability to complete the study protocol
* score high on the IBD knowledge questionnaire (>80%) interventional phase

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-03-10 (Estimated); Study Completion 2022-03-10 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement (PROMIS ) questionnaire | 4 weeks
  Participants will undergo a multiple choice tests with questions relevant to the topic covered. participant will fill the following questioners at base line of the study (before taking the course) and at the end of the study (after 4 weeks). First Questioner out of the 5 is the PROMIS questionnaire:
  Patient-Reported Outcomes Measurement Information System) is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. It can be used with the general population and with individuals living with chronic conditions.
Self-Reported Outcome Measure (SF12) questionnaire | 4 weeks
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.
  The SF-12 uses the same eight domains as the SF-36:
  1. Limitations in physical activities because of health problems.
  2. Limitations in social activities because of physical or emotional problems
  3. Limitations in usual role activities because of physical health problems
  4. Bodily pain
  5. General mental health (psychological distress and well-being)
  6. Limitations in usual role activities because of emotional problems
  7. Vitality (energy and fatigue)
  8. General health perceptions
Lifestyle questionnaire | 4 weeks
  To assess changes within the patients lifestyle. The questioner is designed as open ended questions and multiple choices questions designed to collect relating information to the lifestyle factors including:
  Levels of activity/ Alcohol consumption/ Smoking/ Stress levels/ Diet/
The Medication Adherence Report (MARS-5) questionnaire | 4 weeks
  The Medication Adherence Rating Scale (MARS) The MARS-5 is aimed to collect information regarding patient's level of adherence to the prescribed pharmacological therapy. It is a 5 item scale/ Each item is rated on a 5-point Likert type scale indicating the degree to which the item describes the patient's behavior.
Hospital Anxiety and Depression Scale (HADS) anxiety questionnaire | 4 weeks
  HADS focuses on non-physical symptoms so that it can be used to diagnose depression in people with significant physical ill-health. Any overlap, for instance impaired concentration secondary to pain rather than depression, is usually easy to separate on an individual basis. HADS does not include all of the diagnostic criteria of depression (Diagnostic and Statistical Manual of Mental Disorders, Fourth/Fifth Edition (DSM IV/V)) or all those required by the Health and Work Development Unit (HWDU) National Depression and Long Term Sickness Absence Screening Audit/
  The questionnaire comprises seven questions for anxiety and seven questions for depression

CONTACTS AND LOCATIONS:
Locations (1):
- Sourasky medical center (Ichilov), Tel Aviv, Israel

REFERENCES:
- [Background] Fishman LN, Houtman D, van Groningen J, Arnold J, Ziniel S. Medication knowledge: an initial step in self-management for youth with inflammatory bowel disease. J Pediatr Gastroenterol Nutr. 2011 Dec;53(6):641-5. doi: 10.1097/MPG.0b013e3182285316. PMID 21681113
- [Result] Wardle RA, Mayberry JF. Patient knowledge in inflammatory bowel disease: the Crohn's and Colitis Knowledge Score. Eur J Gastroenterol Hepatol. 2014 Jan;26(1):1-5. doi: 10.1097/MEG.0b013e328365d21a. PMID 24216568
- [Result] Tae CH, Jung SA, Moon HS, Seo JA, Song HK, Moon CM, Kim SE, Shim KN, Jung HK. Importance of Patients' Knowledge of Their Prescribed Medication in Improving Treatment Adherence in Inflammatory Bowel Disease. J Clin Gastroenterol. 2016 Feb;50(2):157-62. doi: 10.1097/MCG.0000000000000431. PMID 26501880
- [Result] Colombara F, Martinato M, Girardin G, Gregori D. Higher levels of knowledge reduce health care costs in patients with inflammatory bowel disease. Inflamm Bowel Dis. 2015 Mar;21(3):615-22. doi: 10.1097/MIB.0000000000000304. PMID 25636120
- [Result] van Groningen J, Ziniel S, Arnold J, Fishman LN. When independent healthcare behaviors develop in adolescents with inflammatory bowel disease. Inflamm Bowel Dis. 2012 Dec;18(12):2310-4. doi: 10.1002/ibd.22937. Epub 2012 Feb 28. PMID 22374585
- [Result] Selinger CP, Eaden J, Selby W, Jones DB, Katelaris P, Chapman G, McDonald C, McLaughlin J, Leong RW, Lal S. Patients' knowledge of pregnancy-related issues in inflammatory bowel disease and validation of a novel assessment tool ('CCPKnow'). Aliment Pharmacol Ther. 2012 Jul;36(1):57-63. doi: 10.1111/j.1365-2036.2012.05130.x. Epub 2012 May 9. PMID 22568682
- [Result] Kim AH, Roberts C, Feagan BG, Banerjee R, Bemelman W, Bodger K, Derieppe M, Dignass A, Driscoll R, Fitzpatrick R, Gaarentstroom-Lunt J, Higgins PD, Kotze PG, Meissner J, O'Connor M, Ran ZH, Siegel CA, Terry H, van Deen WK, van der Woude CJ, Weaver A, Yang SK, Sands BE, Vermeire S, Travis SP. Developing a Standard Set of Patient-Centred Outcomes for Inflammatory Bowel Disease-an International, Cross-disciplinary Consensus. J Crohns Colitis. 2018 Mar 28;12(4):408-418. doi: 10.1093/ecco-jcc/jjx161. PMID 29216349
- [Result] Graff LA, Sexton KA, Walker JR, Clara I, Targownik LE, Bernstein CN. Validating a Measure of Patient Self-efficacy in Disease Self-management Using a Population-based IBD Cohort: The IBD Self-efficacy Scale. Inflamm Bowel Dis. 2016 Sep;22(9):2165-72. doi: 10.1097/MIB.0000000000000856. PMID 27542132
- [Result] Engel T, Ungar B, Ben-Haim G, Levhar N, Eliakim R, Ben-Horin S. Re-phrasing the question: A simple tool for evaluation of adherence to therapy in patients with inflammatory bowel disease. United European Gastroenterol J. 2017 Oct;5(6):880-886. doi: 10.1177/2050640616687838. Epub 2017 Jan 11. PMID 29026602
- [Result] Spiegel BM, Hays RD, Bolus R, Melmed GY, Chang L, Whitman C, Khanna PP, Paz SH, Hays T, Reise S, Khanna D. Corrigendum: development of the NIH Patient-Reported Outcomes Measurement Information System (PROMIS) gastrointestinal symptom scales. Am J Gastroenterol. 2015 Apr;110(4):608. doi: 10.1038/ajg.2015.62. No abstract available. PMID 25853211
- [Result] Eaden JA, Abrams K, Mayberry JF. The Crohn's and Colitis Knowledge Score: a test for measuring patient knowledge in inflammatory bowel disease. Am J Gastroenterol. 1999 Dec;94(12):3560-6. doi: 10.1111/j.1572-0241.1999.01536.x. PMID 10606319